CLINICAL TRIAL: NCT01417676
Title: Pelvic Lymph Node Irradiation With Simultaneous Integrated Boost to Prostate for High Risk Prostate Cancer Patients: A Phase I/II Study
Brief Title: DAPROCA Pelvic Lymph Node Irradiation to Prostate for High Risk Prostate Cancer: Phase I/II Study
Acronym: Propel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Rigshospitalet, Denmark (Other); Herlev Hospital (Other); Odense University Hospital (Other); Vejle Hospital (Other); Aalborg University Hospital (Other); Danish Center for Interventional Research in Radiation Oncology (CIRRO) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIRRO IP080210
Record Dates: First submitted 2011-08-15; First posted 2011-08-16 (Estimated); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; locally advanced; lymph node positive; radiation therapy; morbidity; early morbidity; late morbidity
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients are allocated for lymph node irradiation, either up front combined with prostate irradiation or lymph node irradiation after primary lymph adenectomy after combined with prostate irradiation.
Oversight: Data Monitoring Committee: No

ARMS (1):
- Radiation (Experimental)
  Interventions: Radiation: Radiation: pelvic lymph nodes with boost to prostate

INTERVENTIONS:
Radiation: Radiation: pelvic lymph nodes with boost to prostate — 78(74)Gy/39(37) fractions to prostate, 56(55)GY /39(37) fractions to pelvic lymph nodes, 5 fractions per week.

SUMMARY:
This is a prospective, open label 1 arm study, multicentre, Phase I/II clinical safety study. The trial is designed to gain initial safety and efficacy data on pelvic lymph node radiation with simultaneous integrated boost to prostate in high risk prostate cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* adenocarcinoma
* T3 tumor and either Gleason 8-10 and PSA ≤ 70,or PSA ≥ 30 and PSA ≤ 70, or T1-T3 and PSA ≤ 70 and N1
* no distant metastases

Exclusion Criteria:

* pelvic co-morbidity such as Crohns disease or ulcerative colitis
* uncontrolled heart or lung morbidity
* prior radiation treatment of pelvic region
* age > 75 years

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Incidence of late gastro-intestinal toxicity ≥ grade 2. | 3 years and beyond
  based on CTCAE v.4.0 og in-house questionnaire.

SECONDARY OUTCOMES:
survival | 10 years
recurrence | 10 years
Incidence of late genito-urinary toxicity ≥ grade 2. | 3 years and beyond
  Based on CTCAE vers. 4.0 and in-house questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Lise N Bentzen, MD., Ph.D, Principal Investigator — Aarhus University Hospital, Daproca, CIRRO
Locations (1):
- Dept. of Oncology, Aarhus University Hospital, Aarhus, Denmark